CLINICAL TRIAL: NCT01628250
Title: Clinical Research on the Efficacy and Feasibility of Laparoscopic Complete Mesocolic Excision on Colon Cancer: A Randomized Controlled Study
Brief Title: Laparoscopic Complete Mesocolic Excision on Colon Cancer
Acronym: LCME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Feng (Other)
Responsible Party: Sponsor-Investigator, Bo Feng, Research chair of MIS, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH-MIS
Record Dates: First submitted 2012-06-20; First posted 2012-06-26 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Operation Finding; Complications; Pathology; Quality of Life; Neoplasms Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic complete mesocolic excision (Active Comparator): Randomized group of patients receiving laparoscopic colectomy with the concept of complete mesocolic excision
  Interventions: Procedure: laparoscopic complete mesocolic excision
- D3 laparoscopic colectomy (Active Comparator): Randomized group of patients receiving laparoscopic colectomy with D3-resection
  Interventions: Procedure: D3-laparoscopic colectomy

INTERVENTIONS:
Procedure: laparoscopic complete mesocolic excision — laparoscopic complete mesocolic excision would be applied on randomized group of patients suffering colon cancer and possessing no marked surgical anti-indications. Lap.CME facilitaes medial approach to complete the procedure. CME and HMA are the two arms of the medial approach utilized.
  Other Names: laparoscopic CME; Complete Medial Approach (CMA); Hybrid Medial Approach (HMA)
  Arms: laparoscopic complete mesocolic excision
Procedure: D3-laparoscopic colectomy — D3-laparoscopic colectomy would be applied on randomized group of patients suffering colon cancer and possessing no marked surgical anti-indications.
  Other Names: D3 laparoscopic colectomy
  Arms: D3 laparoscopic colectomy

SUMMARY:
Laparoscopic complete mesocolic excision is a concept that using laparoscopic surgery technique to perform a resection for colon cancer. Besides, the segment of the colon containing the tumor, the resection area should include an intact mesocolon as an envelope to encase the possible route for metastasis. The routes include blood vessels, lymphatic drain and etc. Such hypothesis predicts better histopathological and higher oncological results which turns into better survival rate and better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed colon cancer
* Signed consent

Exclusion Criteria:

* History of malignancy
* Intestinal obstruction or perforation
* Evidence of metastasis by preoperative examinations
* Deformity of spine
* Emergency case
* BMI > 29

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feng, MD/PhD, Principal Investigator — Shanghai Minimally Invasive Surgery Center
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiaotong University school of medicine, Shanghai, Shanghai Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laparoscopic Complete Mesocolic Excision | D3 Laparoscopic Colectomy
Started | 49 | 50
Completed | 49 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Complete Mesocolic Excision | D3 Laparoscopic Colectomy | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 42
  >=65 years | 29 | 28 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 23 | 26 | 49
Region of Enrollment [Number; unit: participants]
  China | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Histopathological Outcomes Obtained Through the Surgeries
Description: number of lymph nodes retrieved
Time Frame: 14 days after the surgery
Measure: Mean (Standard Deviation); unit: nodes
Arm/Group | Laparoscopic Complete Mesocolic Excision | D3 Laparoscopic Colectomy
Number analyzed (Participants) | 49 | 50
nodes | 20.3 (5.8) | 19.2 (6.7)

2. Secondary Outcome: Survival Rate
Description: The follow up to the patients after the surgery to evaluate the oncological results of the technique
Time Frame: 3 years after the surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Laparoscopic Complete Mesocolic Excision | D3 Laparoscopic Colectomy
Serious Adverse Events (participants affected / at risk) | 12/49 | 19/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Complete Mesocolic Excision (N=49) | D3 Laparoscopic Colectomy (N=50)
vessel-related complication (Surgical and medical procedures) | 12 (12) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes